CLINICAL TRIAL: NCT06382974
Title: Evaluation of the Osteoinductivity of Atorvastatin Combined With β-TCP in the Treatment of Bone Defects After Radicular Jaw Cyst Enucleation Using CBCT-based Volumetric Analysis
Brief Title: Evaluation of the Osteoinductivity of Atorvastatin Combined With β-TCP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Yara Gamal Mohamed Mahmoud, post-graduate master student, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3-3-14
Record Dates: First submitted 2024-04-22; First posted 2024-04-25 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Infection; Bone Loss
Keywords: bone regeneration; bone graft; volumetric analysis
MeSH Terms: conditions — Infections; Bone Diseases, Metabolic | interventions — Bone Transplantation

STUDY DESIGN:
Intervention Model Description: A case series study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- bone grafting using atorvastatin combined with beta-TCP (Experimental): the 10 volunteers will undergo cyst enucleation followed by filling the residual bone defects with atorvastatin combined with beta-TCP in the ratio of 0.1 mg: 14 mg.
  Interventions: Procedure: Cyst enucleation and bone grafting

INTERVENTIONS:
Procedure: Cyst enucleation and bone grafting — cyst enucleation followed by bone grafting the residual bone defects using Atorvastatin combined with β-TCP.
  Other Names: Bone grafting

SUMMARY:
This case series study aims to evaluate the local effects of Atorvastatin (which belongs to the family of lipid-lowering drugs, known as statins) combined with β-TCP (which is a synthetic osteoconductive bone graft), on the volume of the residual bone defects and on hastening the bone regeneration after radicular jaw cyst enucleation using CBCT-based volumetric analysis to calculate the shrinkage rate of these defects.

DETAILED DESCRIPTION:
Statement of the problem:

According to the literature, the residual bone defects after medium-large-sized jaw cyst enucleation pose the risk for infection, insufficient healing, and pathological fracture. the gold standard of bone grafting materials remains the autologous bone graft, yet it is accompanied by risks including second surgery, the morbidity of the donor site, excessive bleeding, etc.

Therefore, there is a constant search for alternative bone grafting materials, this is where the addition of atorvastatin to an osteoconductive synthetic bone grafting material (β-TCP) comes in. β-TCP takes anywhere from 6 to 18 months for complete resorption and replacement by bone, according to the literature.

The addition of an osteoinductive material to an osteoconductive grafting material like β-TCP holds two premises; increasing the resorption of the β-TCP particles at the expense of bone deposition, and therefore leads to hastening the bone generation of the residual bone defects.

Rationale:

Studies have shown that the local application of lipid-lowering drugs, statins, induces bone growth by stimulating BMP-2. therefore, the addition of these pharmacological agents to osteoconductive bone graft materials, which lack osteogenic properties, could be a promising approach for bone regeneration.

However, there is still no consensus in the literature on the optimal therapeutic dose and mode of application for statins. Furthermore, limited studies are available in the literature regarding the use of statins especially Atorvastatin as a biological modifier in filling bone defects after cyst enucleation.

Therefore, the purpose of this study is to validate and evaluate the osteoinductivity of statins+ β-TCP combination using the Gouda et al., methodology used in maxillary sinus lifting using simvastatin but instead using atorvastatin in filling the residual defects of medium-large odontogenic radicular cysts (1.5 - 4 cm), which shows the suppressive influence on bone formation, as well as a greater risk for pathological fracture, infection, and insufficient bone healing.

Methodology:

The ratio of atorvastatin to β-TCP will be 0.1 mg: 14 mg, which was the methodology adopted by Gouda et al, based on the methodology of Nyan et al.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients
2. Patients 18 to 40 years old
3. Radicular cyst with a maximum diameter from 1.5 to 4.0 cm;
4. Focal teeth were preserved with root canal treatment;
5. No previous surgical treatment of the cyst site;
6. No evidence of acute inflammation;
7. In good physical status and oral health;
8. Regular attendance at control visits

Exclusion Criteria:

1. Patients < 17 years old
2. Radicular cyst with a maximum diameter < 1.5 cm.
3. Pregnancy or lactation
4. Aggregate systemic pathologies such as diabetes, thyroid disorders, and bone metabolism diseases, among others;
5. Patients taking calcium, bisphosphonates, glucocorticoids, or other drugs that can interfere with the metabolism of bone;
6. Patients with uncontrolled periodontal conditions, endodontic conditions, and other oral disorders;
7. Heavy smokers (10 cigarettes/day or more)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
The Rate of shrinkage of the residual bone defect | 3 moths post-operatively and 6 months post-operatively
  the shrinkage of the residual bone defects after bone grafting, measured from the following formula: pre-operative cyst volume - 3/6 months post-operative defect volume/pre-operative cyst volume x 100%.
  it will be measured radiographically using CBCT through manual segmentation

SECONDARY OUTCOMES:
Incidence of Inflammation at the grafted site | 1 week post-operatively, 3 months post-operatively and 6 months post-operatively
  any signs of inflammation; edema, redness or discharge

CONTACTS AND LOCATIONS:
Overall Officials: Salah Yassin, Study Director — department of oral and maxillofacial surgery, cairo university
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: first in-vivo study to test the methodology adopted in this research — https://pubmed.ncbi.nlm.nih.gov/19397639/
- See also: the clinical study methodology adopted in this research — https://pubmed.ncbi.nlm.nih.gov/28952824/